CLINICAL TRIAL: NCT00273871
Title: A Multi-centre, Randomized, Open-label, Study to Compare Conversion From Calcineurin Inhibitors to Rapamune Versus Standard Therapy in Established Renal Allograft Recipients on Maintenance Therapy With Mild to Moderate Renal Insufficiency.
Brief Title: Study Comparing Conversion From Calcineurin Inhibitors to Rapamune Versus Standard Therapy in Established Renal Allograft Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H1-100535
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2007-05

CONDITIONS: Graft Rejection; Kidney Failure; Kidney Transplantation
Keywords: kidney transplant
MeSH Terms: conditions — Renal Insufficiency | interventions — Cyclosporine; Tacrolimus

INTERVENTIONS:
Drug: Cyclosporin or tacrolimus

SUMMARY:
The purpose of the study is to determine the effect of conversion from calcineurin inhibitor based therapy to Rapamune based therapy in patients with mild to moderate renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Treatment with a calcineurin inhibitor
* Patients with mild to moderate renal insufficiency

Exclusion Criteria:

* Patients with acute rejection
* Patients who received a transplant more than 10 years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 2002-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Difference between treatment groups in renal function at 12 months.

SECONDARY OUTCOMES:
Incidence of acute rejection, patient and graft survival at 12 months, labs and physical examinations, quality of life etc.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For United Kingdom and Ireland, ukmedinfo@wyeth.com